CLINICAL TRIAL: NCT01523340
Title: Phase 4 Study of Response to EGFR-TKI and Correlation With C-met Expression and EGFR Gene Mutation in NSCLC Patients Treated With Erlotinib
Brief Title: A Prospective Observational Study Evaluating c-MET Expression and EGFR Gene Mutation Correlation With Erlotinib Response
Acronym: MENTOR
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Young-Chul Kim, Professor, Chonnam National University Hospital
Other Study IDs: MENTOR_2011
Record Dates: First submitted 2012-01-05; First posted 2012-02-01 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Non-small Cell Lung Cancer Recurrent

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NSCLC tumor tissue for c-MET expression by immuohistochemistry c-MET amplification by silver in situ hybridization EGFR mutation by realtime PCR
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Erlotinib treatment

SUMMARY:
1. Trial design: Prospective observational study
2. Target population: 200 NSCLC patients with histologically or cytologically confirmed stage IV or recurrent NSCLC who have progressive disease after 1st line chemotherapy who consent for study participation and meet the study selection criteria
3. Primary objective: To investigate C-met expression/amplification and EGFR gene mutations in NSCLC patients treated with Erlotinib

   * C-met expression by IHC C-met amplification by SISH EGFR mutation by real time PCR
4. We will also assess the correlation of EGFR mutations and c-MET with clinical outcome (Overall Response Rate, Progression Free survival )
5. Duration of Trial Recruitment: 2 years

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 19~80 year old male or female
* Histologically proven advanced or metastatic NSCLC
* Failed to 1st line chemotherapy
* Tumor tissue for genetic analysis
* Evaluable target lesion by RECIST v1.1
* ECOG performance from 0 to 3
* Expected survival more than 12 weeks

Exclusion Criteria:

* Previous treatment of EGFR-tyrosine kinase inhibitors
* Severe hypersensitivity to erlotinib
* Residual toxicities (above grade 2) after previous chemotherapy
* Total bilirubin more than 1.5x of upper normal limit Liver function tests more than 2.5x of upper normal limits

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed stage IV or recurrent NSCLC who have progressive disease after 1st line chemotherapy who consent for study participation and meet the study selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
The rates of C-met expression/amplification and EGFR gene mutations | Average of 1 year
  To investigate C-met expression/amplification and EGFR gene mutations in NSCLC patients treated with Erlotinib
  : C-met expression by IHC C-met amplification by SISH EGFR mutation by real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, South Korea